CLINICAL TRIAL: NCT05043493
Title: Effect of Platelet Rich Plasma Therapy for Shoulder Osteoarthritis :Double Blinded Randomized Controlled Study
Brief Title: Effect of PRP as Therapy for Shoulder Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ASU 000017585
Record Dates: First submitted 2021-07-18; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-02

CONDITIONS: Shoulder Osteoarthritis
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Injection (study) group (Active Comparator): This group will receive platelet rich plasma (PRP) injection
  Interventions: Procedure: Injection in the intraarticular space of glenohumeral joint
- Control group (Placebo Comparator): This group will receive normal saline (NS) injection
  Interventions: Procedure: Injection in the intraarticular space of glenohumeral joint

INTERVENTIONS:
Procedure: Injection in the intraarticular space of glenohumeral joint — U/S guided injection of platelet rich plasma (PRP) or normal saline (NS)

SUMMARY:
Patients with shoulder osteoarthritis are suffering from pain and disabilities which lead to difficulties in life. The presence of platelet-rich plasma as regenerative therapy which helps in healing of damaged tissues like ligaments and joint might be of great benefit in managing such conditions.

DETAILED DESCRIPTION:
Primary and secondary osteoarthritis of the shoulder occurs due to destruction of the articular surface of the humeral head and glenoid , Patient mainly presented with pain and decreases in the range of motion .

Treatment of shoulder osteoarthritis is often controversial and is typically based on the patient's age, the severity of symptoms, and level of activity, radiographic findings, and medical comorbidities.

The new era of management include regenerative therapy ,Platelet-rich plasma (PRP) is one of the regenerative therapy that prove its effect as injections of a concentration of a patient's own platelets to accelerate the healing of injured tendons, ligaments, muscles and joints.

ELIGIBILITY:
Inclusion Criteria:

* Patient's age: From 21 years.
* Acute symptoms on a background of at least a 3-month history of chronic pain or swelling of the shoulder joint with radiological confirmed (X-ray or MRI)
* Mild or moderate osteoarthritis of the shoulder joint according to The Samilson-Prieto classification.
* Numerical Rating Scale for pain scores greater than five on a 10 scale

Exclusion Criteria:

* Under 21 years of age
* Severe osteoarthritis according to The Samilson-Prieto classification. (Figure 1)
* Neuropsychiatric disorders.
* Immunocompromised patients.
* Active infection or malignancy at the joint.
* Pregnancy and breastfeeding.
* Patients may have thrombocytopenia, bleeding disorders, or on anticoagulant therapy.
* Shoulder surgery within 3 months or inflammatory arthritis; previous infection of the shoulder joint.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Change in patient's pain score | 2 weeks after each injection
  By using NUMERICAL PAIN SCALE patient will mention them pain score on scale from 1 to 10, where the pain score to be included in the study is 5 and more , we will measure pain score for each patient after 2 weeks from injection ,where decrease of the number from the initial recorded number before injection means improvement.

SECONDARY OUTCOMES:
change in the range of motion | 2 weeks after each injection
  This out come will be evaluated by physiotherapist using a device called a goniometer. A goniometer is a metal or plastic handheld device with two arms. Numbers representing angular distance are on the device, The physiotherapist measures the initial angular distance before the injection, and after the injection by 2 weeks Normal range of active movement of the shoulder has been specified by the American Academy of Orthopedic Surgeons (AAOS) to be 180° for flexion and abduction and 90° for external rotation.

OTHER OUTCOMES:
change in the use of analgesic medication | 2 weeks after each injection
  amount of analgesia that needed to inhibit pain, is the patient still in need to pain medication , or he cease it .

CONTACTS AND LOCATIONS:
Overall Officials: Amr Abd Elfatah, proffeseor, Study Director — department of anesthesia ,ICU, and pain management ASU
Locations (1):
- Ainshams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No